CLINICAL TRIAL: NCT03380793
Title: An Open-Lable Multicenter Prospective Non-Randomized Trial to Assess the Efficacy and Safety of Morinidazole With Surgery in Patients With Suppurative or Gangrenous Appendicitis
Brief Title: A Trial to Assess the Efficacy and Safety of Morinidazole in Patients With Appendicitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10090-402
Record Dates: First submitted 2017-11-28; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — morinidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- morinidazole (Experimental): morinidazole and sodium chloride injection (500 mg intravenous, twice daily for 5-7 days) with aztreonam and (or) etimicin.
  Interventions: Drug: morinidazole

INTERVENTIONS:
Drug: morinidazole — morinidazole and sodium chloride injection (500 mg intravenous, twice daily for 5-7 days) with aztreonam and (or) etimicin.

SUMMARY:
To assess the efficacy, safety, tissue distribution of target organ and Population Pharmacokinetic (PPK) of morinidazole and sodium chloride injection with surgery in patients with suppurative or gangrenous appendicitis

DETAILED DESCRIPTION:
Acute appendicitis is among the most common cause of acute abdominal pain. In patients with complicated acute appendicitis, postoperative, broad-spectrum antibiotics are always recommended. Metronidazole, a member of the nitroimidazole drug class, is included in the regimens recommended for improving anaerobic bacteria coverage. The sideeffects of metronidazole include a metallic taste, nausea, transient neutropenia, and peripheral neuropathy. Antimicrobial resistance to metronidazole has emerged after several decades of worldwide use of the drug. Morinidazole, a National Class I Antimicrobial, is a new type of third-generation nitroimidazole antimicrobial that is used for treating amoebiasis, trichomoniasis, and anaerobic bacterial infections, and which exhibits greater activity and less toxicity than metronidazole.

Morinidazole and Sodium Chloride Injection used in pelvic inflammatory disease or appendicitis cases had been approved by CFDA in 2014. This phase 4 study is to assess the efficacy, safety, tissue distribution of target organ and Population Pharmacokinetic (PPK) of morinidazole in patients with suppurative or gangrenous appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 years old
* A diagnosis of suppurative or gangrenous appendicitis based on:

  1. metastatic right lower abdominal pain
  2. lower abdominal tenderness and/or rebound tenderness
  3. pyrexia (axillary temperature ≥ 37.5 °C), a WBC > 10*109/L on routine blood examination
  4. Voluntary signing of written informed consent

Exclusion Criteria:

* patients with an allergy to nitroimidazole
* patients with a history of antibiotic therapy within the last 48 hours
* patients with any condition likely to require broad spectrum antibiotics
* patients who can not evaluate the efficacy or difficult to complete the desired course of treatment
* ALT and / or AST ≥ 1.5 times the ULN, and / or serum creatinine ≥ the ULN
* patients with severe systemic diseases likely to affect therapy (e.g., cardiovascular abnormalities, unstable angina, high blood pressure, severe neuropathy, or epilepsy)
* patients with other diseases or use other drugs which may interfere with the efficacy or safety of the drug
* patients who participated other clinical trials within 6 months before the start of the trial
* Pregnant women, breastfeeding women, women of childbearing age without effective contraceptive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Clinical cure Rate | 5-10 days
  Clinical cure Rate （according to symptoms and signs） at 5-10 days post-therapy

SECONDARY OUTCOMES:
Bacteriological response（Bacterial elimination rate） | 5-10 days
  Bacteriological response (on the first day post-therapy, at 5-10 days post-therapy)
Clinical cure Rate on the first day | the first day
  Clinical cure Rate（according to symptoms and signs）on the first day post-therapy
Tissue distribution | 5-10 days
  Tissue distribution of target organ（Tissue of the appendix）
PPK parameters | 5-10 days
  Area under the plasma concentration versus time curve (AUC) of morinidazole

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, China